CLINICAL TRIAL: NCT05112744
Title: Altération Des Fibres élastiques Dermiques au Cours Des Dermatoses Calcifiantes : étude Structurelle en Microscopie Multiphoton
Brief Title: Alteration of Dermal Elastic Fibers During Calcifying Dermatosis: Structural Study Using Multiphoton Microscopy
Acronym: Calciphoton
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210749
Record Dates: First submitted 2021-10-28; First posted 2021-11-09 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-10

CONDITIONS: Dermatosis
Keywords: Calcified dermatosis; Skin calcifications; Elastic fibres
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The spectrum of pathologies accompanied by tissue mineral deposits is wide. In dermatology, several pathologies are associated with calcium mineral deposits, such as calciphylaxis and pseudoxanthoma elasticum (PXE). However, few studies have been carried out on the chemical characteristics of these deposits, their implication on the pathophysiology and their consequences. This motivated our two previous studies on the characterization of skin mineral deposits during calciphylaxis and sarcoidosis. We have shown that these deposits were most often composed of carbapatite and preferentially localized to elastic fibers. Most calcifying dermatoses are preceded by an inflammatory skin condition. Some authors suspect the digestion of elastin by metalloproteinase (MMP) of the extracellular matrix, thus creating nucleation nuclei favoring phosphocalcic deposits. We thus wish to study the structural alteration of dermal elastic fibers during calcifying dermatoses using multiphoton microscopy, a tool available at the Laboratoire d'Optique et Biosciences (LOB) at the Ecole Polytechnique. Multiphoton microscopy presents several contrast modes that can be used in parallel and without marking. This makes it possible to identify constituent elements of tissues without the use of artificially added fluorescent dyes or proteins, for example fibrillar collagen by the so-called "SHG" contrast and elastin by its intrinsic fluorescence. It is then possible to deeply image an intact tissue, without staining, by specifically visualizing its various components. Used in several studies on the skin, including the LOB, multiphoton microscopy has shown its interest in the characterization of dermal fibers, in particular elastin and collagen fibers, but also in the structural study of these and of their possible alteration. It has thus been applied to the study of skin aging, but also of pathologies leading to degeneration of elastic fibers (PXE) or collagen (Marfan syndrome). The main objective of our project is to characterize the structural alterations of elastic fibers during calcifying dermatoses. The secondary objectives are to study the consequences of skin inflammatory phenomena on the deterioration of elastic fibers and to identify a possible nucleus of phospho-calcium deposits within elastic dermal and vascular fibers. We will thus study human skin biopsies already carried out in the context of the diagnosis of these calcifying dermatoses, skin biopsies from the murine model of PXE and in control, human biopsies of healthy skin from patients of different ages (excision margin of skin tumors). This project should provide a better understanding of the genesis of skin phosphocalcic deposits and provide therapeutic avenues for treating them and limiting their occurrence.

DETAILED DESCRIPTION:
The variety of pathologies accompanied by mineral deposits in tissues is large (cancers, infectious processes, environmental diseases) (1). In dermatology, several pathologies are associated with calcium mineral deposits, such as calciphylaxis and pseudoxanthoma elasticum (PXE). To date, few studies have been carried out on the chemical characteristics of cutaneous mineral deposits, their physiopathological consequences, the occurrence of associated pathologies and their repercussions on human organs.

This has motivated the PhD project of Hester COLBOC, M.D., on the characterization of calcium deposits in various calcifying dermatosis, including calciphylaxis (2) and sarcoidosis (3). This fundamental research project is carried out in the framework of a collaboration between the LCP (Institute of Physico-Chemistry, CNRS, Paris-Saclay University) and AP-HP, in particular in the fields of uro-nephrology (urinary lithiasis) and oncology (4) (calcifications in breast and thyroid cancer). We have shown that skin calcifications consist of carbapatite in calciphylaxis and calcite in sarcoidosis. We have also shown that these deposits are mainly located in the dermal or vessel wall elastic fibres, suggesting a molecular nucleation pathway within these fibers to be explored.

This structural and chemical description is innovative, but does not answer all the questions that arise around these calcium deposits: why do some patients, who present a normal phosphocalcium balance, have massive skin calcifications? Why, on the contrary, do other patients, such as some dialysis patients, present extremely disturbed phosphocalcic balance sheets, but no skin calcification? This paradox raises the possibility of the existence of "nucleation foci" within the elastic dermal and vascular fibers, favouring the precipitation of phosphocalcic deposits in some patients. Some in vitro models have explored these nucleation foci within elastic fibres. (ref Gourgas et al) Quite remarkably, most calcifying dermatosis are preceded by a cutaneous inflammatory state. These skin inflammatory phenomena could also induce the precipitation of calcium deposits. Some authors thus speculate that elastin is digested by metalloproteinase (MMP) in the extracellular matrix, thus creating nucleation foci favouring phosphocalcic deposits. Munavalli et al. showed an increase level of MMP in urinary sample of a patient with calciphylaxis in a context of rapid weight loss (5). They hypothesize that elevated serum MMP levels in this patient could lead to an alteration of the external elastic limit and vascular calcifications. This hypothesis is supported on the other hand by other models of elastic fiber alteration, such as during skin aging (dermatoporosis), in which there is no inflammation and no calcification.

The background hypothesis of our project is that skin inflammation leads to a specific alteration of the elastic fibres, which is conducive to their calcification.

In order to explore this hypothesis, particularly during calciphylaxis and PXE, we propose to use multiphoton microscopy, an imaging technique available at the Laboratoire d'Optique et Biosciences (LOB) at the Ecole Polytechnique. Multiphoton microscopy has been developed in the early 1990s as an alternative to confocal microscopy, to improve in-depth imaging of biological tissues with sub-micrometric resolution. Most importantly, multiphoton microscopy can combine several lodes of contrast in parallel and without any labeling to identify the various elements of a tissue. Second harmonic generation (SHG) signals allow specific imaging of unstained fibrillar collagen with unequalled sensitivity, while two-photon excited fluorescence (2PEF) allows cellular imaging thanks to various intrinsic cellular chromophores as well as elastin imaging in the dermis or in other tissues (see Figure 1) (6).

Multiphoton microscopy has been used in several studies on the skin, including at LOB (see Figure 1), which have proven the high relevance of this technique for the structural characterization of dermal fibers, particularly elastin and collagen fibers, and their possible alteration. It has been applied to the study of skin ageing, as well as to pathologies leading to degeneration of elastic (PXE) or collagen fibres (Marfan Syndrome) (7-9). This technique is therefore highly appropriate for exploring the structure of elastic fibres during cutaneous inflammatory phenomena and calcifying dermatoses.

In parallel, the cutaneous inflammatory process will be explored by other methods. Immuno-histochemistry will be used to detect dermal MMP and X-ray fluorescence (at Synchrotron Soleil, Diffabs line) will be used to evidence intradermal zinc and other metallic deposits, as done in our previous studies (Figure 2).

Figure 2: X-ray fluorescence of a skin biopsy: example of correlation between dermal inflammatory infiltrate (A) and the presence of intradermal Zinc (B), here during a lichenoid reaction on tattoo (images recorded at the Soleil Synchrotron, Diffabs line, by S. Reguer, D. Bazin and H. Colboc).

The main objective of our project is to characterize the structural alterations of elastic fibers during calcifying dermatosis.

The secondary objectives are:

* to study the consequences of cutaneous inflammatory processes on the alteration of elastic fibers,
* to identify a possible nucleation foci for the formation of phospho-calcium deposits within the elastic dermal and vascular fibers.

Skin samples. The study will be mainly performed on human skin, but also on a mouse model of PXE: ABCC6 KO mouse. More precisely, the material studied at LOB will be:

* Human skin biopsies already collected for the diagnosis of these calcifying dermatoses: PXE, calciphylaxis, other calcifying inflammatory dermatoses (lupus panniculitis, dermatomyositis), from the pathology laboratory of the Tenon hospital (Dr Moguelet).
* As controls, human biopsies of healthy skin from patients of different ages, (margin of skin tumour removal), from the Tenon Hospital. We will focuse on patient with advanced skin aging, especially patients with solar elastosis. This model of UV induced elastic fibers alteration is a great control in term of non-inflammatory and non-calcified elastic fibers damages.
* Cutaneous biopsies from the mouse model of PXE (ABCC6 KO mouse) and from matched control mice, from INSERM Unit 1155, Tenon Hospital.

Protocols. All these biopsies will be characterized by multiphoton microscopy by combining 2PEF and SHG contrasts in order to simultaneously image elastic and collagen fibers. In a first step, the experimental protocol will be as follows:

* Production at Tenon Hospital of several serial slides from each biopsy: 1 unstained ("white") slide for multiphoton imaging, 1 slide with usual morphological staining (hematoxylin-eosin-safran, HES), 1 slide with staining highlighting calcium deposits (Von Kossa) and 3 slides with immuno-histochemical labelings of the main MMPs (antibodies against MMP-1, 2 and 9).
* imaging at LOB on a standard brightfield optical microscope (standard and polarized transmitted light, fluorescence, DIC) of all the stained slides over a large field of view by mosaicking; identification of regions of interest (ROI) corresponding to inflammatory processes, tissue remodeling or mineral deposits. Note that mineral deposits are revealed by polarized transmitted light or by phase contrast or DIC.
* X-ray fluorescence imaging at Soleil Synchrotron to identify the metallic deposits present in the biopsies, specially Zinc. This will be done in collaboration with Dominique Bazin (Institute of Physico-Chemistry, CNRS, Paris-Saclay University), which has a strong expertise in mineral imaging in the Diffabs line.
* Multiphoton imaging at LOB of the identified regions of interest, or even on a large field of view by automatically stitching several tiles. Polarization-resolved images will also be carried out in very dense areas or in remodeled areas in order to map the direction of collagen and elastin fibers (10).
* Automated quantitative analysis of multiphoton LOB images to measure several parameters related to the quantity and structure of elastin. Automated quantitative analyses will also be performed on collagen and other structures of interest observed on multiphoton images or histological images. The results of the different imaging modalities will be correlated on each series of slides. Note that automatic analysis is essential both to avoid the usual biases of semi-quantitative analysis and to obtain more informative structural parameters. For instance, the following parameters will be extracted from the elastin images: the mean density of the elastic fibers (per cm², in the papillary dermis and in the reticular dermis), the orientation distribution of the elastic fibers, the entropy and the circular variance of this distribution, the degree of curvature of the elastic fibers, their distance from the mineral deposits.
* Statistical analysis of multimodal data, based on appropriate statistical tests. A priori non-parametric tests (Wilcoxon-Mann-Whitney) will be used in view of the relatively small number of available human samples. A minimum of 8 patients per group will be studied, which should be sufficient due to the accuracy and reproducibility of the automated measurements. If several samples or image series are performed on the same patient, nested statistical tests will be used (nested t-tests or nested Wilcoxon).

In a second step and based on the results of the first step, various items of this protocol will be improved to access more information:

* Multiphoton imaging will be performed in intact murine skin biopsies to better highlight the 3D organization of elastin.
* Advanced fluorescence imaging of inflammation will be performed in ex vivo murine skin, using spectral or FLIM (fluorescence lifetime imaging microscopy) measurements
* Third Harmonic Generation (THG) will be used to visualize the structure of the mineral deposits.

  1. Bazin D, et al. Characterization and some physicochemical aspects of pathological microcalcifications. Chem Rev. 10 oct 2012;112(10):5092-120.

The variety of pathologies accompanied by mineral deposits in tissues is large (cancers, infectious processes, environmental diseases) (1). In dermatology, several pathologies are associated with calcium mineral deposits, such as calciphylaxis and pseudoxanthoma elasticum (PXE). To date, few studies have been carried out on the chemical characteristics of cutaneous mineral deposits, their physiopathological consequences, the occurrence of associated pathologies and their repercussions on human organs.

This has motivated the PhD project of Hester COLBOC, M.D., on the characterization of calcium deposits in various calcifying dermatosis, including calciphylaxis (2) and sarcoidosis (3). This fundamental research project is carried out in the framework of a collaboration between the LCP (Institute of Physico-Chemistry, CNRS, Paris-Saclay University) and AP-HP, in particular in the fields of uro-nephrology (urinary lithiasis) and oncology (4) (calcifications in breast and thyroid cancer). We have shown that skin calcifications consist of carbapatite in calciphylaxis and calcite in sarcoidosis. We have also shown that these deposits are mainly located in the dermal or vessel wall elastic fibres, suggesting a molecular nucleation pathway within these fibers to be explored.

This structural and chemical description is innovative, but does not answer all the questions that arise around these calcium deposits: why do some patients, who present a normal phosphocalcium balance, have massive skin calcifications? Why, on the contrary, do other patients, such as some dialysis patients, present extremely disturbed phosphocalcic balance sheets, but no skin calcification? This paradox raises the possibility of the existence of "nucleation foci" within the elastic dermal and vascular fibers, favouring the precipitation of phosphocalcic deposits in some patients. Some in vitro models have explored these nucleation foci within elastic fibres. (ref Gourgas et al) Quite remarkably, most calcifying dermatosis are preceded by a cutaneous inflammatory state. These skin inflammatory phenomena could also induce the precipitation of calcium deposits. Some authors thus speculate that elastin is digested by metalloproteinase (MMP) in the extracellular matrix, thus creating nucleation foci favouring phosphocalcic deposits. Munavalli et al. showed an increase level of MMP in urinary sample of a patient with calciphylaxis in a context of rapid weight loss (5). They hypothesize that elevated serum MMP levels in this patient could lead to an alteration of the external elastic limit and vascular calcifications. This hypothesis is supported on the other hand by other models of elastic fiber alteration, such as during skin aging (dermatoporosis), in which there is no inflammation and no calcification.

The background hypothesis of our project is that skin inflammation leads to a specific alteration of the elastic fibres, which is conducive to their calcification.

In order to explore this hypothesis, particularly during calciphylaxis and PXE, we propose to use multiphoton microscopy, an imaging technique available at the Laboratoire d'Optique et Biosciences (LOB) at the Ecole Polytechnique. Multiphoton microscopy has been developed in the early 1990s as an alternative to confocal microscopy, to improve in-depth imaging of biological tissues with sub-micrometric resolution. Most importantly, multiphoton microscopy can combine several lodes of contrast in parallel and without any labeling to identify the various elements of a tissue. Second harmonic generation (SHG) signals allow specific imaging of unstained fibrillar collagen with unequalled sensitivity, while two-photon excited fluorescence (2PEF) allows cellular imaging thanks to various intrinsic cellular chromophores as well as elastin imaging in the dermis or in other tissues (see Figure 1) (6).

Multiphoton microscopy has been used in several studies on the skin, including at LOB (see Figure 1), which have proven the high relevance of this technique for the structural characterization of dermal fibers, particularly elastin and collagen fibers, and their possible alteration. It has been applied to the study of skin ageing, as well as to pathologies leading to degeneration of elastic (PXE) or collagen fibres (Marfan Syndrome) (7-9). This technique is therefore highly appropriate for exploring the structure of elastic fibres during cutaneous inflammatory phenomena and calcifying dermatoses.

In parallel, the cutaneous inflammatory process will be explored by other methods. Immuno-histochemistry will be used to detect dermal MMP and X-ray fluorescence (at Synchrotron Soleil, Diffabs line) will be used to evidence intradermal zinc and other metallic deposits, as done in our previous studies (Figure 2).

Figure 2: X-ray fluorescence of a skin biopsy: example of correlation between dermal inflammatory infiltrate (A) and the presence of intradermal Zinc (B), here during a lichenoid reaction on tattoo (images recorded at the Soleil Synchrotron, Diffabs line, by S. Reguer, D. Bazin and H. Colboc).

The main objective of our project is to characterize the structural alterations of elastic fibers during calcifying dermatosis.

The secondary objectives are:

* to study the consequences of cutaneous inflammatory processes on the alteration of elastic fibers,
* to identify a possible nucleation foci for the formation of phospho-calcium deposits within the elastic dermal and vascular fibers.

Skin samples. The study will be mainly performed on human skin, but also on a mouse model of PXE: ABCC6 KO mouse. More precisely, the material studied at LOB will be:

* Human skin biopsies already collected for the diagnosis of these calcifying dermatoses: PXE, calciphylaxis, other calcifying inflammatory dermatoses (lupus panniculitis, dermatomyositis), from the pathology laboratory of the Tenon hospital (Dr Moguelet).
* As controls, human biopsies of healthy skin from patients of different ages, (margin of skin tumour removal), from the Tenon Hospital. We will focuse on patient with advanced skin aging, especially patients with solar elastosis. This model of UV induced elastic fibers alteration is a great control in term of non-inflammatory and non-calcified elastic fibers damages.
* Cutaneous biopsies from the mouse model of PXE (ABCC6 KO mouse) and from matched control mice, from INSERM Unit 1155, Tenon Hospital.

Protocols. All these biopsies will be characterized by multiphoton microscopy by combining 2PEF and SHG contrasts in order to simultaneously image elastic and collagen fibers. In a first step, the experimental protocol will be as follows:

* Production at Tenon Hospital of several serial slides from each biopsy: 1 unstained ("white") slide for multiphoton imaging, 1 slide with usual morphological staining (hematoxylin-eosin-safran, HES), 1 slide with staining highlighting calcium deposits (Von Kossa) and 3 slides with immuno-histochemical labelings of the main MMPs (antibodies against MMP-1, 2 and 9).
* imaging at LOB on a standard brightfield optical microscope (standard and polarized transmitted light, fluorescence, DIC) of all the stained slides over a large field of view by mosaicking; identification of regions of interest (ROI) corresponding to inflammatory processes, tissue remodeling or mineral deposits. Note that mineral deposits are revealed by polarized transmitted light or by phase contrast or DIC.
* X-ray fluorescence imaging at Soleil Synchrotron to identify the metallic deposits present in the biopsies, specially Zinc. This will be done in collaboration with Dominique Bazin (Institute of Physico-Chemistry, CNRS, Paris-Saclay University), which has a strong expertise in mineral imaging in the Diffabs line.
* Multiphoton imaging at LOB of the identified regions of interest, or even on a large field of view by automatically stitching several tiles. Polarization-resolved images will also be carried out in very dense areas or in remodeled areas in order to map the direction of collagen and elastin fibers (10).
* Automated quantitative analysis of multiphoton LOB images to measure several parameters related to the quantity and structure of elastin. Automated quantitative analyses will also be performed on collagen and other structures of interest observed on multiphoton images or histological images. The results of the different imaging modalities will be correlated on each series of slides. Note that automatic analysis is essential both to avoid the usual biases of semi-quantitative analysis and to obtain more informative structural parameters. For instance, the following parameters will be extracted from the elastin images: the mean density of the elastic fibers (per cm², in the papillary dermis and in the reticular dermis), the orientation distribution of the elastic fibers, the entropy and the circular variance of this distribution, the degree of curvature of the elastic fibers, their distance from the mineral deposits.
* Statistical analysis of multimodal data, based on appropriate statistical tests. A priori non-parametric tests (Wilcoxon-Mann-Whitney) will be used in view of the relatively small number of available human samples. A minimum of 8 patients per group will be studied, which should be sufficient due to the accuracy and reproducibility of the automated measurements. If several samples or image series are performed on the same patient, nested statistical tests will be used (nested t-tests or nested Wilcoxon).

In a second step and based on the results of the first step, various items of this protocol will be improved to access more information:

* Multiphoton imaging will be performed in intact murine skin biopsies to better highlight the 3D organization of elastin.
* Advanced fluorescence imaging of inflammation will be performed in ex vivo murine skin, using spectral or FLIM (fluorescence lifetime imaging microscopy) measurements
* Third Harmonic Generation (THG) will be used to visualize the structure of the mineral deposits.

  1. Bazin D, et al. Characterization and some physicochemical aspects of pathological microcalcifications. Chem Rev. 10 oct 2012;112(10):5092-120.
  2. H Colboc, et al. Localization, morphologic features, and chemical composition of calciphylaxis-related skin deposits in patients with calcific uremic arteriolopathy. JAMA Dermatology 2019.
  3. H Colboc, et al. Physicochemical characterization of inorganic deposits associated with granulomas in cutaneous sarcoidosis. Journal of the European Academy of Dermatology and Venereology 2018.
  4. Haka AS, et al. Identifying microcalcifications in benign and malignant breast lesions by probing differences in their chemical composition using Raman spectroscopy. Cancer Res. 15 sept 2002;62(18):5375-80.
  5. Munavalli G, et al. Weight loss-induced calciphylaxis: potential role of matrix metalloproteinases. J Dermatol. 2003;30(12):915-919.
  6. Schanne-Klein M-C. "L'imagerie multiphoton des peaux naturelles et synthétiques. Un nouvel outil pour l'évaluation des produits cosmétiques." Photoniques 88 (2017): 21-24.
  7. Wang, Hequn, et al. "Age-related morphological changes of the dermal matrix in human skin documented in vivo by multiphoton microscopy." Journal of biomedical optics 23.3 (2018): 030501.
  8. Cui, Jason Z., et al. "Quantification of aortic and cutaneous elastin and collagen morphology in Marfan syndrome by multiphoton microscopy." Journal of structural biology 187.3 (2014): 242-253.
  9. Tong, P. L., et al. "A quantitative approach to histopathological dissection of elastin-related disorders using multiphoton microscopy." British Journal of Dermatology 169.4 (2013): 869-879.
  10. G. Ducourthial, J.-S. Affagard, M. Schmeltz, X. Solinas, M. Lopez-Poncelas, C. Bonod-Bidaud, R. Rubio-Amador, F. Ruggiero, J.-M. Allain, E. Beaurepaire, and M.-C. Schanne-Klein, "Monitoring dynamic collagen reorganization during skin stretching with fast polarization-resolved SHG imaging.," J. Biophot. 12, e201800336 (2019).

ELIGIBILITY:
Inclusion Criteria:

* patient with calcified skin disorders
* as controls, patients with skin aging

Exclusion Criteria:

- Patient refusing participation

Ages: 10 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with skin calcified disorders
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-11 (Estimated); Primary Completion 2022-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Characterize structural alteration of the elastic fibers during skin diseases associated to ectopic calcifications | One year

SECONDARY OUTCOMES:
Identify a potential nucleation foci for phospho-calcium deposits within dermal and vascular elastic fibers. | One year

CONTACTS AND LOCATIONS:
Overall Officials: Hester Colboc, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Service de gériatrie plaies et cicatrisation, Paris, France

IPD SHARING:
Plan to Share IPD: No